CLINICAL TRIAL: NCT03962777
Title: Efficacy of Oil Pulling Therapy With Coconut Oil on Four Day Supragingival Plaque Growth: a Randomized Crossover Clinical Trial
Brief Title: Efficacy of Oil Pulling Therapy on Supragingival Plaque Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, asistant professor, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BaskentU5
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Gingivitis
Keywords: gingivitis; oil pulling
MeSH Terms: conditions — Gingivitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oil pulling (Experimental): patients used oil pulling therapy for 4 days
  Interventions: Other: oil pulling
- chlorhexidine (Active Comparator): patients used chlorhexidine digluconate for 4 days
  Interventions: Other: chlorhexidine

INTERVENTIONS:
Other: chlorhexidine — patients used chx moutrinses for four days
  Arms: chlorhexidine
Other: oil pulling — patients used oil pulling for four days
  Arms: oil pulling

SUMMARY:
Oil pulling is a method based on Ayurvedic medicine which aims to obtain local and systemic benefits by swirling oils in the oral cavity for a period of 15 minutes, before spitting it out.12 Although the exact mechanism of action is not clear, there are some proposed theories. One proposed theory is the saponification or "soap making" process which occurs as a result of alkali hydrolysis of fat.9 Second theory speculates the inhibition of plaque formation and adhesion of bacteria due to the viscous nature of the oil. 13 According to the third theory, presence of antioxidants in oil prevent lipid peroxidation and thus help to the destruction of microorganisms and potentiating the action of Vitamin E in the oral cavity.14 The effect of oil pulling on halitosis and the use of oil pulling in addition to conventional oral hygiene practices was investigated in some studies13,15,16 but to the best knowledge of the authors, no study has evaluated the plaque-inhibiting effects of oil pulling. Therefore this study was conducted to evaluate the plaque-inhibiting effects of oil pulling using 4- day plaque regrowth study model17,18 compared to 0.2% CHX-containing mouthrinse. The tested hypothesis was that oil pulling would perform plaque regrowth inhibition as well as the CHX-containing mouthrinse.

DETAILED DESCRIPTION:
The study was a single-center, observer masked, cross-over design with subjects randomly allocated to treatment sequences. During a 2-week preparatory period, participants rendered plaque, calculus and stain free by a thorough scaling and polishing of the teeth by both hand and ultrasonic instruments and were instructed in self-performed plaque control. At the end of the preparatory period, all subjects had clinically healthy gingiva.

Participants were randomly allocated to two groups by closed envelop system (BM) and masked to the mouthrinse received. The tested products and regimens of use are shown in Table 1. Mouthrinses were filled in identical but coded bottles. Instructions for usage was written on the bottles. On day 1 (Monday) of each study periods, after disclosing the teeth with erythrosine all subjects received scaling and polishing to remove plaque and extrinsic stain and disclosing of the teeth was repeated. By this way it was confirmed that all participants had a plaque score of 0 at baseline. Subjects were then asked to refrain from all forms of tooth cleaning and to apply the rinsing regimen. The tested agents included the following: 1) 0.2 % chlorhexidine mouthrinse ( 10 mL, twice daily for 30 seconds) 2) Coconut oil (10 Ml, twice daily 15-20 minute) All agents were to be used after breakfast and dinner and the subjects should be avoided rinsing, eating and drinking during the first hour after rinsing. During the 4- day period, the use of any other rinse, chewing gum or toothpaste was not allowed. The mouthrinses were in identical bottles but total subject blindness cannot be possible due to the taste, color, consistency, rinsing time differences.

On day 5 (Friday), subjects received an oral soft tissue examination and were asked to complete a standardized questionnaire to evaluate their attitudes with regard to the product used. The patients were asked about the flavor of the mouthrinse, the alteration in the taste of food and drinks, the perception of the plaque reduction, the staining that the mouthrinse created, the feeling to create nausea. After the completion of the questionnaire, each subject was scored for staining using Lobene stain index.19 After that, disclosing was performed with erythrosine and plaque scoring was performed using the Turesky et al. 20 modification of the Quigley and Hein index.21 Stain and plaque indices were recorded from the buccal and lingual surfaces of all fully erupted permanent teeth, with the exception of the third molars. In addition, Gingival Index (GI) and bleeding on probing (bop) were recorded from six sites of each teeth. All clinical examinations were performed by a single clinician (YS) who was masked to the study.

After recording the clinical parameters, subjects received a polishing to remove all plaque and tooth stain if present and 14 days of washout periods were allowed after 4- day period. 22 During the wash out period, the subjects returned to normal oral hygiene methods with a standard toothbrush* and a fluoride containing tooth paste**. These procedures were repeated until each participant used each of the rinses.

ELIGIBILITY:
Inclusion Criteria:

* no systemic disease
* having ≥ 22 natural teeth,
* having no removable or fixed prostheses or fixed and removable orthodontic appliances.

Exclusion criteria:

* use of antibiotics and anti-inflammatory drugs in previous 6 months;
* allergy to any ingredient used in the study;
* smokers;
* pregnant of lactating females;
* history of mouthrinses, gels or chewing gums use that contains antimicrobial agents in the preceding 3 months
* having teeth with probing depth ≥4mm and signs of gingival inflammation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
plaque index | day 4
  plaque regrowth inhibition will be tested using the Turesky et al. 21 modification of the Quigley and Hein index.a score of 0 to 5 is assigned to each facial and lingual nonrestored surface of all the teeth except third molars, as follows: 0: No plaque; 1:Separate flecks of plaque at the cervical margin of the tooth; 2:A thin continuos band of plaque (up to one mm) at the cervical margin of the tooth; 3: A band of plaque wider than one mm but covering less than one-third of the crown of the tooth; 4:Plaque covering at least one-third but less than two-thirds of the crown of the tooth; 5: Plaque covering two-thirds or more of the crown of the tooth. An index for the entire mouth is determined by dividing the total score by the number surfaces ( a maximum of 2 x 2 x 14 = 56 surfaces) examined.lower values means that the agent has better plaque inhbiting effect

CONTACTS AND LOCATIONS:
Overall Officials: yasemin sezgin, asst prof, Study Director — başkent university, faculty of dentistry
Locations (1):
- Yasemin Sezgin, Ankara, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No